CLINICAL TRIAL: NCT03278613
Title: Neuromodulation for Accidental Bowel Leakage
Acronym: NOTABLe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NICHD Pelvic Floor Disorders Network (Network)
Collaborators: University of Alabama at Birmingham (Other); University of California, San Diego (Other); Duke University (Other); Women and Infants Hospital of Rhode Island (Other); RTI International (Other); University of Pennsylvania (Other); University of Pittsburgh (Other); Kaiser Permanente (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12865-29; 2U24HD069031-06 (NIH); 2UG1HD069013-06 (NIH); 5UG1HD041267-18 (NIH); 5UG1HD069010-07 (NIH); 5UG1HD069006-07 (NIH); 5UG1HD041261-17 (NIH); 5UG1HD054214-12 (NIH); 5UG1HD054241-12 (NIH)
Record Dates: First submitted 2017-09-06; First posted 2017-09-11 (Actual); Results first posted 2021-05-14 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Fecal Incontinence; Bowel Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will remain masked to subject treatment assignment throughout the trial. To maintain masking of participants, the duration of treatment sessions for both the PTNS and sham groups will be 30 minutes and will be conducted with subjects in a supine position with the knees comfortably abducted and flexed. The leg and foot involved in treatment will be obscured from the subject's view with a portable anesthesia drape frame to which an exam sheet will be secured.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Percutaneous Tibial Nerve Stimulation (PTNS) (Experimental): PTNS treatment entails insertion of a 36 gauge needle electrode at a 60 degree angle 3-4 cm deep towards the tibial nerve, approximately 5 cm or 3 finger breadths cephalad to the medial malleolus and posterior to the tibia. The PTNS grounding electrode, placed near the calcaneus and the needle electrode will be connected to the ES-130 device pulse generator.
  Interventions: Device: ES-130
- Validated Sham (Sham Comparator): Sham treatment will use the Streitberger acupuncture placebo needle in the same location as the needle electrode for PTNS. The sham uses an active gel surface electrode pad placed on the bottom of the foot just below the fifth (smallest) toe. This location is not part of the acupuncture nerve pathway connected to the bladder, pelvis or any major organs. Electrical current is delivered to this pad via a TENS unit resulting in sensory stimulation.
  Interventions: Device: ES-130

INTERVENTIONS:
Device: ES-130 — The ES-130 device will be used for the indication of "Posterior Tibial Nerve Stimulation for the treatment of fecal incontinence" using the FDA-approved protocol for treatment of urge urinary incontinence (UUI) in the PFDN NOTABLe study. There is no PTNS device cleared by the FDA for the indication of FI treatment; therefore, this is considered an investigational device.

SUMMARY:
This study is a multi-center, randomized clinical trial of women with refractory accidental bowel leakage (ABL) symptoms who have failed to achieve satisfactory symptom control from 2 first-line treatments for ABL: supervised pelvic muscle training (PMT) and constipating medication. The purpose of this study is to compare percutaneous tibial nerve stimulation (PTNS) to a validated sham to determine if PTNS is effective for the treatment of fecal incontinence (FI) in women.

The investigators will test the null hypothesis that change from baseline in St. Mark's (Vaizey) score after 12 weeks of stimulation is not significantly different in women with symptomatic ABL receiving PTNS treatments compared to women receiving sham PTNS treatments.

DETAILED DESCRIPTION:
The overarching goal of this randomized clinical trial is to determine if PTNS is more effective than sham PTNS for the treatment of FI in women after 12 weeks of treatment and 1 year after initiating treatment. This is a two-part trial with a Run-In Phase prior to randomization. The trial has the following primary aim:

To determine whether the change from baseline in St. Mark's (Vaizey) score in women with symptomatic ABL undergoing PTNS differs from sham after 12 weeks of stimulation.

Additional secondary aims include:

1. To compare changes from baseline in self-reported functional outcomes after 12 weekly stimulation sessions in both PTNS and sham groups in Part 1.
2. To determine whether symptom relief amongst study "responders" can be sustained for one year with maintenance treatments in Part II.
3. To determine the impact of completing a bowel diary and receiving education on FI on symptom severity.
4. To determine the ability of the PFDN ABL phone app bowel diary to detect changes from baseline in fecal incontinence episodes recorded to after 12 weeks of stimulation sessions.
5. To determine the association between St. Mark's score and both fat and fiber intake alone and in combination.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years of age
* FI symptoms ≥ 3 months
* Baseline St. Mark's score of ≥ 12
* Attended ≥ 2 supervised PMT for ABL
* Intolerance, unwillingness, or inadequate response to constipating medications
* Current negative colon cancer screening based on the USPSTF's recommendation for colorectal cancer screening (2016)

Exclusion Criteria:

* Previous PTNS treatment
* History of uncontrolled diarrhea in the past 3 months (usual or most common stool type over the preceding 3 months of 7 on the Bristol Stool Form Scale)
* History of severe constipation in the past 3 months (usual or most common stool type over the preceding 3 months of 1 on the Bristol Stool Form Scale)
* History of inflammatory bowel disease (includes Crohn's disease and ulcerative colitis, but does not include irritable bowel disease)
* Unrepaired rectovaginal fistula/chronic 4th degree laceration
* Full thickness rectal prolapse
* History of congenital anorectal malformation
* History of bowel resection surgery for any indication
* Minor anal procedures within 6 months for treatment of ABL (injection of bulking agent or radiofrequency energy) or ligation of hemorrhoids
* Prior pelvic or abdominal radiation
* Diagnosis of cancer of the descending colon or anus
* Diagnosis of cancer in the region where the PTNS or sham needles or surface electrodes would be placed
* Pacemaker, implantable defibrillator
* Current use of Interstim sacral nerve stimulator or TENS in the pelvic region, back, or legs
* Clinically significant neurological disorders known to affect anal continence
* Coagulopathy
* Severe peripheral edema preventing accurate placement of PTNS needles
* Chronic swollen, infected, inflamed skin or skin eruptions (e.g., phlebitis, thrombophlebitis, varicose veins) in the region where the PTNS or sham needles or surface electrodes would be placed
* Metal implant in foot/toes near TENS electrode location
* Marked sensory deficit (numbness) of feet or ankles in the region where the PTNS or sham needles or surface electrodes would be placed
* Childbirth within the last 3 months
* Pregnant or planning to become pregnant during the study duration 1 year; a urine pregnancy test will be performed and must be negative by the first intervention visit if the participant is of childbearing potential
* Unwilling to use acceptable form of contraceptive if the participant is of childbearing potential
* Participation in another intervention trial impacting bowel function
* Inability to provide informed consent, complete questionnaires independently, or to attend intervention sessions
* Unable or unwilling to complete the bowel diary in Run-In Phase (valid diary defined as data from ≥ 10 of 14 days with minimum of 3 consecutive days per week)
* Unwilling to download bowel diary app onto smartphone if the participant owns a smartphone
* Visual impairment prohibiting reading the paper diary, the smart phone screen
* Unable to speak, read, or write in English or Spanish at a basic level

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Halina M Zyczynski, MD, Study Chair — Magee-Women's Hospital, Department of Obstetrics and Gynecology
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Kaiser Permanente -- Downey, Downey, California
  - University of California at San Diego, UCSD Women's Pelvic Medicine Center, La Jolla, California
  - Kaiser Permanente -- San Diego, San Diego, California
  - Duke University, Duke Division of Urogynecology and Reconstructive Pelvic Surgery, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Magee-Women's Hospital, Department of Obstetrics and Gynecology, Pittsburgh, Pennsylvania
  - Brown/ Women and Infants Hospital of Rhode Island, Center for Women's Pelvic Medicine and Reconstructive Surgery, Providence, Rhode Island
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zyczynski HM, Richter HE, Sung VW, Lukacz ES, Arya LA, Rahn DD, Visco AG, Mazloomdoost D, Carper B, Gantz MG; NICHD Pelvic Floor Disorders Network. Percutaneous Tibial Nerve Stimulation vs Sham Stimulation for Fecal Incontinence in Women: NeurOmodulaTion for Accidental Bowel Leakage Randomized Clinical Trial. Am J Gastroenterol. 2022 Apr 1;117(4):654-667. doi: 10.14309/ajg.0000000000001605. PMID 35354778
- [Derived] Zyczynski HM, Arya LA, Lukacz ES, Richter HE, Rahn DD, Sung VW, Visco AG, Shaffer A, Jelovsek JE, Rogers R, Mazloomdoost D, Gantz MG; Eunice Kennedy Shriver NICHD Pelvic Floor Disorders Network (PFDN). Design of a Randomized Controlled Trial of Percutaneous Posterior Tibial Nerve Stimulation for the Treatment of Refractory Fecal Incontinence in Women: The NeurOmodulaTion for Accidental Bowel Leakage Study. Female Pelvic Med Reconstr Surg. 2021 Dec 1;27(12):726-734. doi: 10.1097/SPV.0000000000001050. PMID 33950027

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Percutaneous Tibial Nerve Stimulation (PTNS) | Validated Sham
Started | 111 | 55
Completed | 108 | 54
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- PTNS: PTNS treatment entails insertion of a 36 gauge needle electrode at a 60 degree angle 3-4 cm deep towards the tibial nerve, approximately 5 cm or 3 finger breadths cephalad to the medial malleolus and posterior to the tibia. The PTNS grounding electrode, placed near the calcaneus and the needle electrode will be connected to the ES-130 device pulse generator.
  ES-130: The ES-130 device will be used for the indication of "Posterior Tibial Nerve Stimulation for the treatment of fecal incontinence" using the FDA-approved protocol for treatment of urge urinary incontinence (UUI) in the PFDN NOTABLe study. There is no PTNS device cleared by the FDA for the indication of FI treatment; therefore, this is considered an investigational device.
- Sham: Sham treatment will use the Streitberger acupuncture placebo needle in the same location as the needle electrode for PTNS. The sham uses an active gel surface electrode pad placed on the bottom of the foot just below the fifth (smallest) toe. This location is not part of the acupuncture nerve pathway connected to the bladder, pelvis or any major organs. Electrical current is delivered to this pad via a TENS unit resulting in sensory stimulation.
  ES-130: The ES-130 device will be used for the indication of "Posterior Tibial Nerve Stimulation for the treatment of fecal incontinence" using the FDA-approved protocol for treatment of urge urinary incontinence (UUI) in the PFDN NOTABLe study. There is no PTNS device cleared by the FDA for the indication of FI treatment; therefore, this is considered an investigational device.
- Total: Total of all reporting groups
Arm/Group | PTNS | Sham | Total
Number analyzed (Participants) | 111 | 55 | 166
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (12) | 63.8 (11) | 63.6 (12)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 111 | 55 | 166
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 6 | 16
  Not Hispanic or Latino | 99 | 49 | 148
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 10 | 9 | 19
  White | 95 | 39 | 134
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 7
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.2 (7) | 29.7 (6) | 29.4 (7)
Current Smoker [Count of Participants; unit: Participants]
  Yes | 9 | 5 | 14
  No | 102 | 50 | 152
Ever Pregnant [Count of Participants; unit: Participants]
  Yes | 107 | 50 | 157
  No | 4 | 5 | 9
Number of Vaginal Deliveries [Median (Full Range); unit: deliveries per participant] | 2 [0 to 9] | 2 [0 to 7] | 2 [0 to 9]
Number of Cesarean Deliveries [Median (Full Range); unit: deliveries per participant] | 0 [0 to 4] | 0 [0 to 1] | 0 [0 to 4]
Menstrual Status [Count of Participants; unit: Participants]
  pre-menopausal | 11 | 4 | 15
  post-menopausal | 92 | 49 | 141
  not sure | 8 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline St. Mark's (Vaizey) Score
Description: The primary outcome measure is the change from baseline in St. Mark's (Vaizey) Score 12 weeks after treatment initiation to compare the outcomes of post-tibial nerve stimulation (PTNS) versus sham stimulation. The St. Mark's (Vaizey) score, published in 1999, is commonly used in clinical studies and reports and was based on the Jorge-Wexner score but added two further items for assessment: the use of constipating medication and the presence of fecal urgency. Minimum score is 0 = perfect continence; maximum score is 24 = totally incontinent. Change from baseline is calculated as Week [4, 8, or 12] Score minus the score at baseline.
Time Frame: 4, 8, and 12 Weeks
Population: An intent-to-treat (ITT) analysis which included all eligible participants who were randomized and who provided outcome data after baseline was performed.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 108 | 54
units on a scale
  Week 4: number analyzed (Participants) | 102 | 50
  Week 4 | -2.8 [-3.5 to -2] | -3.3 [-4.5 to -2.1]
  Week 8: number analyzed (Participants) | 105 | 52
  Week 8 | -4.3 [-5.2 to -3.3] | -4.1 [-5.4 to -2.9]
  Week 12: number analyzed (Participants) | 104 | 54
  Week 12 | -5.3 [-6.3 to -4.3] | -3.9 [-5.3 to -2.6]

2. Secondary Outcome: Responder to Treatment
Description: Responder status is based on the primary chnage from St. Mark's Score. A responder is defined as any particpant with at least a 4 point reduction in score compared to their baseline score
Time Frame: 4, 8, and 12 Weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 108 | 54
Participants
  Week 4: number analyzed (Participants) | 102 | 50
  Week 4: Responder | 39 | 24
  Week 4: Non-responder | 63 | 26
  Week 8: number analyzed (Participants) | 105 | 52
  Week 8: Responder | 54 | 29
  Week 8: Non-responder | 51 | 23
  Week 12: number analyzed (Participants) | 104 | 54
  Week 12: Responder | 64 | 26
  Week 12: Non-responder | 40 | 28

3. Secondary Outcome: Change From Baseline Number of Fecal Incontinence Events Per Week
Description: Based on data collected from participant-completed diaries at baseline, 8, and 12 weeks, the outcome variable is computed as the difference in number of fecal incontinence episodes per week at 8 and 12 weeks and the number of fecal incontinence episodes at baseline.
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: episodes per week
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 106 | 53
episodes per week
  Week 8: number analyzed (Participants) | 103 | 52
  Week 8 | -2.4 [-3.1 to -1.6] | -1.6 [-3.2 to 0]
  Week 12: number analyzed (Participants) | 101 | 51
  Week 12 | -2.3 [-3.2 to -1.5] | -2.1 [-3.7 to -0.4]

4. Secondary Outcome: Change From Baseline Number of Urge Fecal Incontinence Events Per Week
Description: Based on data collected from participant-completed diaries at baseline, 8, and 12 weeks, the outcome variable is computed as the difference in number of urge fecal incontinence episodes per week at 8 and 12 weeks and the number of urge fecal incontinence episodes at baseline.
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: episodes per week
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 106 | 53
episodes per week
  Week 8: number analyzed (Participants) | 103 | 52
  Week 8 | -1.3 [-1.8 to -0.8] | -0.4 [-1.1 to 0.2]
  Week 12: number analyzed (Participants) | 101 | 51
  Week 12 | -1.1 [-1.6 to -0.6] | -0.8 [-1.4 to -0.1]

5. Secondary Outcome: Change From Baseline Number of Bowel Movements Per Week
Description: Based on data collected from participant-completed diaries at baseline, 8, and 12 weeks, the outcome variable is computed as the difference in number of bowel movements per week at 8 and 12 weeks and the number of bowel movements at baseline.
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: episodes per week
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 106 | 53
episodes per week
  Week 8: number analyzed (Participants) | 103 | 52
  Week 8 | -1.8 [-3 to -0.6] | -0.2 [-1.6 to 1.1]
  Week 12: number analyzed (Participants) | 101 | 51
  Week 12 | -1.8 [-2.8 to -0.9] | -1.5 [-2.8 to -0.2]

6. Secondary Outcome: Change From Baseline Number of Urge Bowel Movements Per Week
Description: Based on data collected from participant-completed diaries at baseline, 8, and 12 weeks, the outcome variable is computed as the difference in number of urge bowel movements per week at 8 and 12 weeks and the number of urge bowel movements at baseline.
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: episodes per week
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 106 | 53
episodes per week
  Week 8: number analyzed (Participants) | 103 | 52
  Week 8 | -1.9 [-2.9 to -0.8] | -1.1 [-2.2 to -0.1]
  Week 12: number analyzed (Participants) | 101 | 51
  Week 12 | -2.3 [-3.2 to -1.3] | -2.2 [-3.3 to -1.1]

7. Secondary Outcome: Change From Baseline Number of Days Without Fecal Incontinence Episodes Per Week
Description: Based on data collected from participant-completed diaries at baseline, 8, and 12 weeks, the outcome variable is computed as the difference in number of days without fecal incontinence episodes per week at 8 and 12 weeks and the number of days without fecal incontinence episodes at baseline.
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: episodes per week
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 106 | 53
episodes per week
  Week 8: number analyzed (Participants) | 103 | 52
  Week 8 | 1 [0.6 to 1.4] | 0.8 [0.3 to 1.3]
  Week 12: number analyzed (Participants) | 101 | 51
  Week 12 | 1.3 [0.9 to 1.7] | 0.8 [0.2 to 1.4]

8. Secondary Outcome: 50% Improvement in Fecal Incontinence Episodes Per Week
Description: Based on data collected from participant-completed diaries at baseline, 8, and 12 weeks, the outcome is calculated as any participant with a 50% reduction in fecal incontinence episodes per week at 8 and 12 weeks compared to the fecal incontinence episodes at baseline
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 102 | 50
Participants
  Week 8: number analyzed (Participants) | 99 | 49
  Week 8: >= 50% Improvement | 38 | 14
  Week 8: < 50% Improvement | 61 | 35
  Week 12: number analyzed (Participants) | 97 | 48
  Week 12: >= 50% Improvement | 51 | 19
  Week 12: < 50% Improvement | 46 | 29

9. Secondary Outcome: 75% Improvement in Fecal Incontinence Episodes Per Week
Description: Based on data collected from participant-completed diaries at baseline, 8, and 12 weeks, the outcome is calculated as any participant with a 75% reduction in fecal incontinence episodes per week at 8, and 12 weeks compared to the fecal incontinence episodes at baseline.
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 102 | 50
Participants
  Week 8: number analyzed (Participants) | 99 | 49
  Week 8: >= 75% Improvement | 19 | 10
  Week 8: < 75% Improvement | 80 | 39
  Week 12: number analyzed (Participants) | 97 | 48
  Week 12: >= 75% Improvement | 32 | 13
  Week 12: < 75% Improvement | 65 | 35

10. Secondary Outcome: Patient Global Impression-Improvement
Description: The Patient Global Impression of Improvement (PGI-I) is a patient-reported measure of perceived improvement with treatment, as assessed on a scale of 1 (very much better) to 7 (very much worse). Included here are participants who had improvement as indicated by a rating of 1 (very much better) or 2 (much better)
Time Frame: 4, 8, and 12 Weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 108 | 54
Participants
  Week 4: number analyzed (Participants) | 103 | 50
  Week 4: Improved | 20 | 13
  Week 4: No improvement | 83 | 37
  Week 8: number analyzed (Participants) | 106 | 50
  Week 8: Improved | 36 | 17
  Week 8: No improvement | 70 | 33
  Week 12: number analyzed (Participants) | 103 | 54
  Week 12: Improved | 47 | 21
  Week 12: No improvement | 56 | 33

11. Other Pre Specified Outcome: Change From Baseline ABLe Liquid Score
Description: The ABLE Liquid Score is a subscale of the validated Accidental Bowel Leakage Evaluation (ABLE) questionnaire which assesses the impact and severity of the leakage of liquid stool. Minimum score is 0 = no problem with liquid stool leakage; maximum score is 4 = frequent, bothersome leakage of large amounts of liquid stool. Change from baseline is calculated as Week [8 or 12] Score minus the score at baseline.
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 106 | 54
units on a scale
  Week 8: number analyzed (Participants) | 106 | 51
  Week 8 | -0.3 [-0.4 to -0.1] | -0.5 [-0.8 to -0.2]
  Week 12: number analyzed (Participants) | 103 | 54
  Week 12 | -0.6 [-0.8 to -0.4] | -0.7 [-1 to -0.4]

12. Other Pre Specified Outcome: Change From Baseline ABLe Solid Score
Description: The ABLE Solid Score is a subscale of the validated Accidental Bowel Leakage Evaluation (ABLE) questionnaire which assesses the impact and severity of the leakage of solid stool. Minimum score is 0 = no problem with solid stool leakage; maximum score is 4 = frequent, bothersome leakage of large amounts of solid stool. Change from baseline is calculated as Week [8 or 12] Score minus the score at baseline.
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 106 | 54
units on a scale
  Week 8: number analyzed (Participants) | 106 | 51
  Week 8 | -0.5 [-0.7 to -0.3] | -0.4 [-0.6 to -0.1]
  Week 12: number analyzed (Participants) | 103 | 54
  Week 12 | -0.7 [-0.9 to -0.5] | -0.7 [-1 to -0.4]

13. Other Pre Specified Outcome: Change From Baseline ABLe Mucus Score
Description: The ABLE Mucus Score is a subscale of the validated Accidental Bowel Leakage Evaluation (ABLE) questionnaire which assesses the impact and severity of the leakage of mucus from the rectum. Minimum score is 0 = no problem with mucus leakage from the rectum; maximum score is 4 = frequent, bothersome leakage of large amounts of mucus from the rectum. Change from baseline is calculated as Week [8 or 12] Score minus the score at baseline.
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 105 | 54
units on a scale
  Week 8: number analyzed (Participants) | 104 | 51
  Week 8 | -0.5 [-0.7 to -0.3] | -0.4 [-0.7 to -0.1]
  Week 12: number analyzed (Participants) | 102 | 54
  Week 12 | -0.7 [-0.9 to -0.5] | -0.4 [-0.7 to -0.1]

14. Other Pre Specified Outcome: Change From Baseline ABLe Gas Score
Description: The ABLE Gas Score is a subscale of the validated Accidental Bowel Leakage Evaluation (ABLE) questionnaire which assesses the impact and severity of the leakage of gas from the rectum. Minimum score is 0 = no problem with gas leakage from the rectum; maximum score is 4 = frequent and bothersome leakage of gas from the rectum. Change from baseline is calculated as Week [8 or 12] Score minus the score at baseline.
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 106 | 54
units on a scale
  Week 8: number analyzed (Participants) | 106 | 51
  Week 8 | -0.3 [-0.5 to -0.1] | -0.2 [-0.5 to 0.1]
  Week 12: number analyzed (Participants) | 103 | 54
  Week 12 | -0.4 [-0.6 to -0.3] | -0.4 [-0.7 to -0.1]

15. Other Pre Specified Outcome: Change From Baseline ABLe Predictability/Awareness Score
Description: The ABLE Predictability/Awareness Score is a subscale of the validated Accidental Bowel Leakage Evaluation (ABLE) questionnaire which assesses the predictability of bowel leakage events. Minimum score is 0 = no problems with leakage; maximum score is 4 = leakage without awareness or predictability. Change from baseline is calculated as Week [8 or 12] Score minus the score at baseline.
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 106 | 54
units on a scale
  Week 8: number analyzed (Participants) | 106 | 51
  Week 8 | 0 [-0.2 to 0.1] | 0 [-0.2 to 0.2]
  Week 12: number analyzed (Participants) | 103 | 54
  Week 12 | -0.2 [-0.4 to -0.1] | 0 [-0.2 to 0.2]

16. Other Pre Specified Outcome: Change From Baseline ABLe Control Score
Description: The ABLE Control Score is a subscale of the validated Accidental Bowel Leakage Evaluation (ABLE) questionnaire which assesses the ability to control bowel movements. Minimum score is 0 = no problems with urgency to empty bowels wthout warning; maximum score is 4 = frequent and bothersome urgency to empty bowels wthout warning.
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 106 | 54
units on a scale
  Week 8: number analyzed (Participants) | 106 | 51
  Week 8 | -0.3 [-0.5 to -0.2] | -0.3 [-0.6 to -0.1]
  Week 12: number analyzed (Participants) | 103 | 54
  Week 12 | -0.6 [-0.8 to -0.4] | -0.6 [-0.9 to -0.3]

17. Other Pre Specified Outcome: Change From Baseline ABLe Ancillary Bowel Symptoms Score
Description: The ABLE Ancillary Bowel Symptoms Score is a subscale of the validated Accidental Bowel Leakage Evaluation (ABLE) questionnaire which assesses the frequency and impact of ancially bowel symptoms. Minimum score is 0 = no problems with pain or incomplete emptying; maximum score is 4 = frequent and bothersome pain or incomplete emptying.
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 106 | 54
units on a scale
  Week 8: number analyzed (Participants) | 106 | 51
  Week 8 | -0.4 [-0.5 to -0.2] | -0.3 [-0.6 to -0.1]
  Week 12: number analyzed (Participants) | 103 | 54
  Week 12 | -0.7 [-0.9 to -0.5] | -0.4 [-0.6 to -0.1]

18. Other Pre Specified Outcome: Change From Baseline ABLe Overall Score
Description: The ABLE Overall Score is the summary score of the validated Accidental Bowel Leakage Evaluation (ABLE) questionnaire which assesses the frequency and impact of accidental bowel leakage and related symptoms. Minimum score is 0 = no problems with bowel leakage and related symptoms; maximum score is 4 = frequent and bothersome problems with bowel leakage and related symptoms.
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 106 | 54
units on a scale
  Week 8: number analyzed (Participants) | 106 | 51
  Week 8 | -0.4 [-0.5 to -0.2] | -0.3 [-0.6 to -0.1]
  Week 12: number analyzed (Participants) | 103 | 54
  Week 12 | -0.7 [-0.9 to -0.5] | -0.4 [-0.6 to -0.1]

19. Other Pre Specified Outcome: Patient Global Symptom Control
Description: The Patient Global Symptom Control (PGSC) is a patient-reported measure of perceived agreement that symptoms are under control, as assessed on a scale of 1 (Disagree Strongly) to 5 (Agree Strongly). Included here are participants who had reported disagreements as indicated by a rating of 1 (Disagree Strongly) or 2 (Disagree)
Time Frame: Baseline and 4, 8, and 12 Weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 111 | 55
Participants
  Baseline: number analyzed (Participants) | 111 | 54
  Baseline: No Control | 18 | 10
  Baseline: Control | 93 | 44
  Week 4: number analyzed (Participants) | 105 | 50
  Week 4: No Control | 46 | 25
  Week 4: Control | 59 | 25
  Week 8: number analyzed (Participants) | 106 | 52
  Week 8: No Control | 70 | 33
  Week 8: Control | 36 | 19
  Week 12: number analyzed (Participants) | 104 | 54
  Week 12: No Control | 82 | 40
  Week 12: Control | 22 | 14

20. Other Pre Specified Outcome: Change From Baseline FIQL Lifestyle Score
Description: The FIQL Lifestyle Score is a subscale of the validated Fecal Incontinence Quality of Life (FIQL) questionnaire which assesses the impact of accidental bowel leakage on quality of life. Minimum score is 1 = lower functional quality of life; maximum score is 5 = higher functional quality of life. Change from baseline is calculated as Week [8 or 12] Score minus the score at baseline.
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 106 | 54
units on a scale
  Week 8: number analyzed (Participants) | 105 | 51
  Week 8 | 0.3 [0.2 to 0.5] | 0.4 [0.2 to 0.6]
  Week 12: number analyzed (Participants) | 102 | 54
  Week 12 | 0.6 [0.5 to 0.8] | 0.4 [0.2 to 0.6]

21. Other Pre Specified Outcome: Change From Baseline FIQL Coping Score
Description: The FIQL Coping Score is a subscale of the validated Fecal Incontinence Quality of Life (FIQL) questionnaire which assesses the impact of accidental bowel leakage on quality of life. Minimum score is 1 = lower functional quality of life; maximum score is 5 = higher functional quality of life. Change from baseline is calculated as Week [8 or 12] Score minus the score at baseline.
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 106 | 54
units on a scale
  Week 8: number analyzed (Participants) | 106 | 51
  Week 8 | 0.4 [0.3 to 0.5] | 0.4 [0.2 to 0.6]
  Week 12: number analyzed (Participants) | 102 | 54
  Week 12 | 0.6 [0.5 to 0.8] | 0.5 [0.3 to 0.7]

22. Other Pre Specified Outcome: Change From Baseline FIQL Depression Score
Description: The FIQL Depression Score is a subscale of the validated Fecal Incontinence Quality of Life (FIQL) questionnaire which assesses the impact of accidental bowel leakage on quality of life. Minimum score is 1 = lower functional quality of life; maximum score is 5 = higher functional quality of life. Change from baseline is calculated as Week [8 or 12] Score minus the score at baseline.
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 106 | 54
units on a scale
  Week 8: number analyzed (Participants) | 106 | 51
  Week 8 | 0.3 [0.2 to 0.4] | 0.2 [0 to 0.4]
  Week 12: number analyzed (Participants) | 102 | 54
  Week 12 | 0.5 [0.4 to 0.6] | 0.2 [0.1 to 0.4]

23. Other Pre Specified Outcome: Change From Baseline FIQL Embarrassment Score
Description: The FIQL Embarrassment Score is a subscale of the validated Fecal Incontinence Quality of Life (FIQL) questionnaire which assesses the impact of accidental bowel leakage on quality of life. Minimum score is 1 = lower functional quality of life; maximum score is 5 = higher functional quality of life. Change from baseline is calculated as Week [8 or 12] Score minus the score at baseline.
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 106 | 54
units on a scale
  Week 8: number analyzed (Participants) | 105 | 51
  Week 8 | 0.4 [0.3 to 0.5] | 0.4 [0.2 to 0.6]
  Week 12: number analyzed (Participants) | 102 | 53
  Week 12 | 0.7 [0.6 to 0.9] | 0.4 [0.3 to 0.6]

24. Other Pre Specified Outcome: Change From Baseline FISI Patient Score
Description: The FISI Patient Score is a summary score of the validated Fecal Incontinence Severity Index questionnaire which provides a summary metric of the severity of fecal incontinence from the patient's perspective. Minimum score is 0 = no fecal incontinence; maximum score is 61 = very severe fecal incontinence. Change from baseline is calculated as Week [8 or 12] Score minus the score at baseline.
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 102 | 53
units on a scale
  Week 8: number analyzed (Participants) | 100 | 50
  Week 8 | -4.9 [-7.1 to -2.8] | -5.9 [-8.7 to -3.1]
  Week 12: number analyzed (Participants) | 95 | 52
  Week 12 | -7.5 [-9.7 to -5.3] | -6.7 [-10.1 to -3.3]

25. Other Pre Specified Outcome: Change From Baseline FISI Doctor Score
Description: The FISI Doctor Score is a summary score of the validated Fecal Incontinence Severity Index questionnaire which provides a summary metric of the severity of fecal incontinence from the doctor's perspective. Minimum score is 0 = no fecal incontinence; maximum score is 57 = very severe fecal incontinence. Change from baseline is calculated as Week [8 or 12] Score minus the score at baseline.
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 102 | 53
units on a scale
  Week 8: number analyzed (Participants) | 100 | 50
  Week 8 | -5 [-7.3 to -2.8] | -6.3 [-9.2 to -3.4]
  Week 12: number analyzed (Participants) | 95 | 52
  Week 12 | -7.4 [-9.8 to -5] | -7 [-10.5 to -3.5]

26. Other Pre Specified Outcome: Change From Baseline MMHQ Incontinence Impact Score
Description: The MMHQ Incontinence Impact Score is a subscale of the validated Modified-Manchester Health questionnaire (MMHq) which provides a health-related quality of life rating. Minimum score is 0 = high quality of life; maximum score is 100 = low quality of life. Change from baseline is calculated as Week [8 or 12] Score minus the score at baseline.
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 106 | 54
units on a scale
  Week 8: number analyzed (Participants) | 104 | 51
  Week 8 | -9.4 [-14.5 to -4.2] | -11.3 [-17.9 to -4.6]
  Week 12: number analyzed (Participants) | 103 | 52
  Week 12 | -17.2 [-23 to -11.5] | -15.9 [-23.4 to -8.3]

27. Other Pre Specified Outcome: Change From Baseline MMHQ Role Limitations Score
Description: The MMHQ Role Limitations Score is a subscale of the validated Modified-Manchester Health questionnaire (MMHq) which provides a health-related quality of life rating. Minimum score is 0 = high quality of life; maximum score is 100 = low quality of life. Change from baseline is calculated as Week [8 or 12] Score minus the score at baseline.
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 104 | 53
units on a scale
  Week 8: number analyzed (Participants) | 103 | 49
  Week 8 | -9.8 [-14.6 to -5.1] | -3.1 [-10.4 to 4.3]
  Week 12: number analyzed (Participants) | 101 | 52
  Week 12 | -17.5 [-22.6 to -12.3] | -9.9 [-17.1 to -2.6]

28. Other Pre Specified Outcome: Change From Baseline MMHQ Physical Limitations Score
Description: The MMHQ Physical Limitations Score is a subscale of the validated Modified-Manchester Health questionnaire (MMHq) which provides a health-related quality of life rating. Minimum score is 0 = high quality of life; maximum score is 100 = low quality of life. Change from baseline is calculated as Week [8 or 12] Score minus the score at baseline.
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 104 | 53
units on a scale
  Week 8: number analyzed (Participants) | 102 | 49
  Week 8 | -10.3 [-15.3 to -5.3] | -3.8 [-9.2 to 1.6]
  Week 12: number analyzed (Participants) | 100 | 52
  Week 12 | -20.4 [-25.5 to -15.2] | -10.6 [-16.6 to -4.5]

29. Other Pre Specified Outcome: Change From Baseline MMHQ Social Limitations Score
Description: The MMHQ Social Limitations Score is a subscale of the validated Modified-Manchester Health questionnaire (MMHq) which provides a health-related quality of life rating. Minimum score is 0 = high quality of life; maximum score is 100 = low quality of life. Change from baseline is calculated as Week [8 or 12] Score minus the score at baseline.
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 106 | 54
units on a scale
  Week 8: number analyzed (Participants) | 102 | 50
  Week 8 | -9.6 [-15.3 to -3.9] | -1.8 [-7.5 to 3.9]
  Week 12: number analyzed (Participants) | 102 | 53
  Week 12 | -14.8 [-20.1 to -9.5] | -8.6 [-14.6 to -2.7]

30. Other Pre Specified Outcome: Change From Baseline MMHQ Personal Relationship Score
Description: The MMHQ Personal Relationship Score is a subscale of the validated Modified-Manchester Health questionnaire (MMHq) which provides a health-related quality of life rating. Minimum score is 0 = high quality of life; maximum score is 100 = low quality of life. Change from baseline is calculated as Week [8 or 12] Score minus the score at baseline.
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 75 | 35
units on a scale
  Week 8: number analyzed (Participants) | 70 | 28
  Week 8 | -5 [-11.6 to 1.6] | -2.2 [-11.5 to 7]
  Week 12: number analyzed (Participants) | 71 | 35
  Week 12 | -6.2 [-11.3 to -1] | -11.4 [-23.2 to 0.4]

31. Other Pre Specified Outcome: Change From Baseline MMHQ Emotional Function Score
Description: The MMHQ Emotional Function Score is a subscale of the validated Modified-Manchester Health questionnaire (MMHq) which provides a health-related quality of life rating. Minimum score is 0 = high quality of life; maximum score is 100 = low quality of life. Change from baseline is calculated as Week [8 or 12] Score minus the score at baseline.
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 104 | 54
units on a scale
  Week 8: number analyzed (Participants) | 103 | 51
  Week 8 | -7.2 [-11.7 to -2.7] | -4.6 [-10.6 to 1.5]
  Week 12: number analyzed (Participants) | 101 | 52
  Week 12 | -14.4 [-19.1 to -9.6] | -7.4 [-14.3 to -0.4]

32. Other Pre Specified Outcome: Change From Baseline MMHQ Sleep/Energy Score
Description: The MMHQ Sleep/Energy Score is a subscale of the validated Modified-Manchester Health questionnaire (MMHq) which provides a health-related quality of life rating. Minimum score is 0 = high quality of life; maximum score is 100 = low quality of life. Change from baseline is calculated as Week [8 or 12] Score minus the score at baseline.
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 104 | 53
units on a scale
  Week 8: number analyzed (Participants) | 101 | 50
  Week 8 | -7.2 [-11.4 to -3] | -4.3 [-10.8 to 2.3]
  Week 12: number analyzed (Participants) | 98 | 51
  Week 12 | -11 [-15.2 to -6.8] | -6.4 [-12.4 to -0.3]

33. Other Pre Specified Outcome: Change From Baseline MMHQ Severity Measures Score
Description: The MMHQ Severity Measures Score is a subscale of the validated Modified-Manchester Health questionnaire (MMHq) which provides a health-related quality of life rating. Minimum score is 0 = high quality of life; maximum score is 100 = low quality of life. Change from baseline is calculated as Week [8 or 12] Score minus the score at baseline.
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 105 | 51
units on a scale
  Week 8: number analyzed (Participants) | 104 | 47
  Week 8 | -9.1 [-13.2 to -5] | -10.7 [-15.9 to -5.6]
  Week 12: number analyzed (Participants) | 101 | 50
  Week 12 | -17 [-21.3 to -12.6] | -11.8 [-17 to -6.6]

34. Other Pre Specified Outcome: Change From Baseline CRAIQ Score
Description: The Pelvic Floor Impact Questionnaire short form (PFIQ-7) measuring the impact of bladder, bowel, and vaginal symptoms on a woman's daily activities, relationships and emotions is composed of 3 scales of 7 questions each: the Urinary Impact Questionnaire (UIQ; range 0-100), the Pelvic Organ Prolapse Impact Questionnaire (POPIQ; range 0-100), and the Colorectal-Anal Impact Questionnaire (CRAIQ; range 0-100). Scores are calculated by multiplying the mean value of all answered questions for a scale by 100 divided by 3. The range of responses is: 0-100 with 0 (least negative impact) to 100 (most negative impact). Change = (Week [8, 12] Score - Baseline Score). Lower scores indicate better function / fewer symptoms.
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 106 | 54
units on a scale
  Week 8: number analyzed (Participants) | 105 | 51
  Week 8 | -12.9 [-17.1 to -8.7] | -12.8 [-19.6 to -5.9]
  Week 12: number analyzed (Participants) | 103 | 54
  Week 12 | -19.1 [-24.2 to -14] | -14.5 [-22.2 to -6.9]

35. Other Pre Specified Outcome: Change From Baseline POPIQ Score
Description: as for outcome 34
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 106 | 54
units on a scale
  Week 8: number analyzed (Participants) | 105 | 51
  Week 8 | -3.3 [-7.2 to 0.7] | -5.1 [-8.8 to -1.5]
  Week 12: number analyzed (Participants) | 103 | 54
  Week 12 | -5.2 [-8.1 to -2.3] | -5.6 [-9.8 to -1.4]

36. Other Pre Specified Outcome: Change From Baseline UIQ Score
Description: as for outcome 34
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 106 | 54
units on a scale
  Week 8: number analyzed (Participants) | 105 | 51
  Week 8 | -3.3 [-6.4 to -0.1] | -10.2 [-15.3 to -5]
  Week 12: number analyzed (Participants) | 103 | 54
  Week 12 | -7.2 [-10.6 to -3.8] | -10.5 [-16.5 to -4.6]

37. Other Pre Specified Outcome: Change From Baseline PFIQ Score
Description: as for outcome 34
Time Frame: 8 and 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 106 | 54
units on a scale
  Week 8: number analyzed (Participants) | 105 | 51
  Week 8 | -19.4 [-27.7 to -11.1] | -28.1 [-39.9 to -16.2]
  Week 12: number analyzed (Participants) | 103 | 54
  Week 12 | -31.5 [-40.3 to -22.7] | -30.7 [-43.7 to -17.6]

38. Other Pre Specified Outcome: Change From Baseline PAC-SYM Abdominal Score
Description: The Patient Assessment of Constipation - Symptom (PAC-SYM) ia a validated form measuring the frequency and severity of chronic constipation. It consists of an overall score (range: 0-4) consisting of 3 subscales across 12 question: the Abdominal score (range 0-4), the Rectal Score (range 0-4), and the Stool Score (range 0-4). Scores are calculated as the mean of non-mising responses. The range of responses is: 0-4 with 0 (Absent) to 4 (Very sever). Change = (Week 12 Score - Baseline Score). Lower scores indicate less severe constipation.
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 103 | 53
units on a scale | -0.4 [-0.6 to -0.3] | -0.2 [-0.4 to 0]

39. Other Pre Specified Outcome: Change From Baseline PAC-SYM Rectal Score
Description: as for outcome 38
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 103 | 54
units on a scale | -0.1 [-0.3 to 0.0] | -0.1 [-0.3 to 0.1]

40. Other Pre Specified Outcome: Change From Baseline PAC-SYM Stool Score
Description: as for outcome 38
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 103 | 54
units on a scale | -0.3 [-0.5 to -0.1] | -0.2 [-0.5 to 0.0]

41. Other Pre Specified Outcome: Change From Baseline PAC-SYM Total Score
Description: The Patient Assessment of Constipation - Symptom (PAC-SYM) is a validated form measuring the frequency and severity of chronic constipation. It consists of an overall score (range: 0-4) consisting of 3 subscales across 12 question: the Abdominal score (range 0-4), the Rectal Score (range 0-4), and the Stool Score (range 0-4). Scores are calculated as the mean of non-missing responses. The range of responses is: 0-4 with 0 (Absent) to 4 (Very severe). Change = (Week 12 Score - Baseline Score). Lower scores indicate less severe constipation.
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 103 | 54
units on a scale | -0.3 [-0.4 to -0.2] | -0.2 [-0.4 to 0.0]

42. Other Pre Specified Outcome: Change From Baseline PISQ-IR NSA-PR Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised measures the impact of incontinence symptoms on sexual function and satisfaction. The Not Sexually Active-Partner Related (NSA-PR) ranges from 1 to 4 with higher scores indicating greater sexual function. The outcome is calculated as the difference in score at 12 weeks and the score at baseline.
Time Frame: 12 Weeks
Population: An intent-to-treat (ITT) analysis which included all eligible participants who were randomized and who provided outcome data after baseline was performed. This measure was only collected from participants that were not sexually active.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 43 | 29
units on a scale | 0.1 [-0.3 to 0.4] | -0.1 [-0.4 to 0.1]

43. Other Pre Specified Outcome: Change From Baseline PISQ-IR NSA-CS Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised measures the impact of incontinence symptoms on sexual function and satisfaction. The Not Sexually Active-Condition Specific (NSA-CS) ranges from 1 to 4 with higher scores indicating greater sexual function. The outcome is calculated as the difference in score at 12 weeks and the score at baseline.
Time Frame: 12 Weeks
Population: as for outcome 42
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 40 | 29
units on a scale | 0.2 [-0.1 to 0.5] | 0.2 [-0.2 to 0.6]

44. Other Pre Specified Outcome: Change From Baseline PISQ-IR NSA-GQA Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised measures the impact of incontinence symptoms on sexual function and satisfaction. The Not Sexually Active-Global Quality Rating (NSA-GQA) ranges from 1 to 4.5 with higher scores indicating greater sexual function. The outcome is calculated as the difference in score at 12 weeks and the score at baseline.
Time Frame: 12 Weeks
Population: as for outcome 42
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 41 | 28
units on a scale | 0.4 [0.1 to 0.6] | 0.3 [0 to 0.5]

45. Other Pre Specified Outcome: Change From Baseline PISQ-IR NSA-CI Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised measures the impact of incontinence symptoms on sexual function and satisfaction. The Not Sexually Active-Condition Impact (NSA-CI) ranges from 1 to 4 with higher scores indicating greater sexual function. The outcome is calculated as the difference in score at 12 weeks and the score at baseline.
Time Frame: 12 Weeks
Population: An intent-to-treat (ITT) analysis which included all eligible participants who were randomized and who provided outcome data after baseline was performed. This measure was only collected for participants that were not sexually active.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 40 | 28
units on a scale | 0.4 [0.1 to 0.7] | 0.3 [0.0 to 0.6]

46. Other Pre Specified Outcome: Change From Baseline PISQ-IR SA-AO Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised measures the impact of incontinence symptoms on sexual function and satisfaction. The Sexually Active-Arousal Orgasm (SA-AO) ranges from 1 to 5 with higher scores indicating greater sexual function. The outcome is calculated as the difference in score at 12 weeks and the score at baseline.
Time Frame: 12 Weeks
Population: An intent-to-treat (ITT) analysis which included all eligible participants who were randomized and who provided outcome data after baseline was performed. This measure is only calculated for participants that were sexually active.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 46 | 21
units on a scale | 0.2 [0.1 to 0.4] | 0.2 [0.0 to 0.4]

47. Other Pre Specified Outcome: Change From Baseline PISQ-IR SA-PR Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised measures the impact of incontinence symptoms on sexual function and satisfaction. The Sexually Active-Partner Related (SA-PR) ranges from 1 to 4 with higher scores indicating greater sexual function. The outcome is calculated as the difference in score at 12 weeks and the score at baseline.
Time Frame: 12 Weeks
Population: An intent-to-treat (ITT) analysis which included all eligible participants who were randomized and who provided outcome data after baseline was performed. This measure is only collected from participants that were sexually active.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 44 | 19
units on a scale | 0.1 [0.0 to 0.3] | 0.0 [-0.2 to 0.2]

48. Other Pre Specified Outcome: Change From Baseline PISQ-IR SA-CS Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised measures the impact of incontinence symptoms on sexual function and satisfaction. The Sexually Active-Condition Specific (SA-CS) ranges from 1 to 5 with higher scores indicating greater sexual function. The outcome is calculated as the difference in score at 12 weeks and the score at baseline.
Time Frame: 12 Weeks
Population: An intent-to-treat (ITT) analysis which included all eligible participants who were randomized and who provided outcome data after baseline was performed. This measure was only collected from participants that were sexually active.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 45 | 20
units on a scale | 0.3 [0.1 to 0.6] | 0.5 [0.2 to 0.8]

49. Other Pre Specified Outcome: Change From Baseline PISQ-IR SA-GQR Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised measures the impact of incontinence symptoms on sexual function and satisfaction. The Sexually Active-Global Quality Rating (SA-GQR) ranges from 1 to 4.75 with higher scores indicating greater sexual function. The outcome is calculated as the difference in score at 12 weeks and the score at baseline.
Time Frame: 12 Weeks
Population: as for outcome 48
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 46 | 21
units on a scale | 0.3 [0.1 to 0.6] | 0.4 [-0.1 to 0.9]

50. Other Pre Specified Outcome: Change From Baseline PISQ-IR SA-CI Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised measures the impact of incontinence symptoms on sexual function and satisfaction. The Sexually Active-Condition Impact (SA-CI) ranges from 1 to 4 with higher scores indicating greater sexual function. The outcome is calculated as the difference in score at 12 weeks and the score at baseline.
Time Frame: 12 Weeks
Population: as for outcome 48
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 46 | 21
units on a scale | 0.4 [0.2 to 0.6] | 0.3 [0.0 to 0.6]

51. Other Pre Specified Outcome: Change From Baseline PISQ-IR SA-D Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised measures the impact of incontinence symptoms on sexual function and satisfaction. The Sexually Active-Desire (SA-D) ranges from 1 to 5 with higher scores indicating greater sexual function. The outcome is calculated as the difference in score at 12 weeks and the score at baseline.
Time Frame: 12 Weeks
Population: as for outcome 48
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 45 | 21
units on a scale | 0.0 [-0.1 to 0.2] | 0.2 [-0.2 to 0.6]

52. Other Pre Specified Outcome: Change From Baseline PISQ-IR SA-AVG Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised measures the impact of incontinence symptoms on sexual function and satisfaction. The Sexually Active-Average (SA-AVG) ranges from 1 to 5 with higher scores indicating greater sexual function. The outcome is calculated as the difference in score at 12 weeks and the score at baseline.
Time Frame: 12 Weeks
Population: as for outcome 48
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 44 | 19
units on a scale | 0.2 [0.1 to 0.4] | 0.3 [0.1 to 0.5]

53. Other Pre Specified Outcome: Change From Baseline FIAI Hygiene Index Score
Description: The Fecal Incontinence Adaptation Index (FIAI) is a validated form which measures the adaptation behavios resulting from fecal incontinence. It consists of two subscales: Hygiene (range: 0-100) and Avoidance (range: 0-100). Scores are cal calculated as the average of the non-missing responses multiplied by 25. The outcome is calculated as the difference in score at 12 weeks and the score at baseline.
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 101 | 54
units on a scale | -10.2 [-14 to -6.5] | -2.8 [-8.4 to 2.9]

54. Other Pre Specified Outcome: Change From Baseline FIAI Avoidance Index Score
Description: as for outcome 53
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 101 | 54
units on a scale | -12.8 [-16.1 to -9.4] | -6.4 [-12.2 to -0.6]

55. Other Pre Specified Outcome: Change From Baseline SF-12 Aggregate Physical Score
Description: The 12-Item Short-Form Health Survey (SF-12) is a validated survey which assesses overall physical and mental health. The Aggregate Physical Score ranges from 24 to 56.6 with higher scores indicating greater physical health. The outcome is calculated as the difference in score at 12 weeks and the score at baseline.
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 89 | 50
units on a scale | 2.6 [1.1 to 4.2] | 2.1 [-1 to 5.3]

56. Other Pre Specified Outcome: Change From Baseline SF-12 Aggregate Mental Score
Description: The 12-Item Short-Form Health Survey (SF-12) is a validated survey which assesses overall physical and mental health. The Aggregate Mental Score ranges from 19.06 to 60.86 with higher scores indicating greater mental health. The outcome is calculated as the difference in score at 12 weeks and the score at baseline
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PTNS | Sham
Number analyzed (Participants) | 89 | 50
units on a scale | 0.9 [-1.3 to 3.1] | -0.7 [-4.2 to 2.9]

ADVERSE EVENTS:
Time Frame: 12 Weeks
Arm/Group | PTNS | Sham
All-Cause Mortality (participants affected / at risk) | 1/111 | 0/55
Serious Adverse Events (participants affected / at risk) | 4/111 | 2/55
Other Adverse Events (participants affected / at risk) | 72/111 | 30/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PTNS (N=111) | Sham (N=55)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PTNS (N=111) | Sham (N=55)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Chalazion (Eye disorders) | 1 (1) | 0 (0)
Photopsia (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2)
Anal paraesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (6) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 6 (9) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0)
Application site pain (General disorders) | 2 (2) | 0 (0)
Application site paraesthesia (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 2 (2) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Medical device site haemorrhage (General disorders) | 9 (14) | 0 (0)
Medical device site pain (General disorders) | 1 (1) | 0 (0)
Puncture site pain (General disorders) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Multiple allergies (Immune system disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 4 (4) | 1 (1)
Eye infection (Infections and infestations) | 2 (2) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 7 (8) | 2 (2)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 3 (3) | 1 (1)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 14 (14) | 4 (4)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 6 (7) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Colonoscopy (Investigations) | 1 (1) | 0 (0)
Endoscopy gastrointestinal (Investigations) | 1 (1) | 0 (0)
Oesophagogastroduodenoscopy (Investigations) | 1 (1) | 0 (0)
Gluten sensitivity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (7) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 11 (16) | 2 (2)
Sciatica (Nervous system disorders) | 2 (2) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Urge incontinence (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Fibrocystic breast disease (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal pain (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Abdominal hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Abdominoplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Medical device removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-07-03): https://cdn.clinicaltrials.gov/large-docs/13/NCT03278613/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-28): https://cdn.clinicaltrials.gov/large-docs/13/NCT03278613/SAP_001.pdf
  • Informed Consent Form (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/13/NCT03278613/ICF_002.pdf